CLINICAL TRIAL: NCT05058326
Title: Severity of Fecal Incontinence and Manometric Values Using the Anopress® Device in Women
Acronym: MANOPRESS
Status: Completed | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Other Study IDs: 052020
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Fecal Incontinence; Anal; Sphincter, Incontinence; Incontinence, Urge
Keywords: Anal manometry; Anal portable manometry; Fecal incontinence severity; Endoanal ultrasound
MeSH Terms: conditions — Fecal Incontinence; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEST GROUP: Women with fecal incontinence referred to outpatients clinic.
  Interventions: Diagnostic Test: Portable endoanal manometry; Diagnostic Test: Endoanal ultrasound; Other: Incontinence severity scale questionaires

INTERVENTIONS:
Diagnostic Test: Portable endoanal manometry — Endoanal manometry values will be obtained using de Anopress® device. Fecal incontinence severity questionaries will be filled and collected.
Diagnostic Test: Endoanal ultrasound — To assess the integrity of the anal canal.
Other: Incontinence severity scale questionaires — Wexner and St. Mark's scales.

SUMMARY:
The purpose of this study is to stablish a correlation between fecal incontinence severity scales (Wexner & St. Mark's) and manometric values obtained using the Anopress® portable manometry and values obtained using endoanal ultrasound in women with fecal incontinence.

DETAILED DESCRIPTION:
The Anopress® portable anal manometry will be used to measure the pressures of the anal canal in different phases: rest, squeeze, strain and endurance.

All female patients referred with the diagnosis of fecal incontinence giving written informed consent will undergo a endoanal portable manometry at our outpatients clinics. They will be asked to fill out the severity questionaries (Sant Mark's and Wexner). All data will be collected for analysis.

An endoanal ultrasound will be performed in all patients to assess the sphincter integrity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of fecal incontinence
* Age ≥ 18 years.
* Informed consent signed by the patient and the researcher.

Exclusion Criteria:

* Patients with psychiatric illnesses, addictions or any disorder that prevents understanding of the study.
* Inability to read or understand the questionnaires.
* Inability to read or understand any of the informed consent languages (Catalan, Spanish).
* Any patient who, due to his medical characteristics, presents a high individual risk when being included and completing the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years referred to our outpatient's clinic with the clinical diagnosis of fecal incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Stablish a correlation between Wexner fecal incontinence severity scales and manometric values obtained using the Anopress® portable manometry in women with fecal incontinence | During the procedure
  Spearman and Pearson correlation will be used to assess correlations between values
Stablish a correlation between St. Mark's fecal incontinence severity scales and manometric values obtained using the Anopress® portable manometry in women with fecal incontinence | During the procedure
  Spearman and Pearson correlation will be used to assess correlations between values

SECONDARY OUTCOMES:
Stablish a correlation between St.Mark's fecal incontinence severity scales and values obtained using endoanal ultrasound in women with fecal incontinence | During the procedure
  Spearman and Pearson correlation will be used to assess correlations between values
Stablish a correlation between Wexner fecal incontinence severity scales and values obtained using endoanal ultrasound in women with fecal incontinence | During the procedure
  Spearman and Pearson correlation will be used to assess correlations between values

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No